CLINICAL TRIAL: NCT02692183
Title: Mapping Functional Networks of Brain Activity (Brain Network Activation, BNA) Based on Analysis of Evoked Response Potential (ERP) Signals in Patients With Essential Tremor or Parkinson Disease Before and After MR-guided Focused Ultrasound (FUS) Thalamotomy for Tremor
Brief Title: Mapping Functional Networks of Brain Activity Using EEG in Patients With Essential Tremor or Parkinson Disease Before and After MR-guided Focused Ultrasound Thalamotomy for Tremor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: ElMindA Ltd (Industry); InSightec (Industry)
Responsible Party: Sponsor
Other Study IDs: SHEBA-SH-2805-15-CTIL
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson Disease-tremor; Essential Tremor
Keywords: Parkinson's disease; ET; EEG; FUS; BNA; Essential tremor
MeSH Terms: conditions — Essential Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson Disease (PD) tremor patients: Patients with PD before and after MRI guided Focused ultrasound thalamotomy
- Essential tremor (ET) patients: Patients with ET before and after MRIFocused ultrasound guided thalamotomy

SUMMARY:
A cornerstone in PD and ET research is the investigation of neurophysiological changes as potential bio-markers that could help in tracking disease progression and response to therapy. Electroencephalography (EEG) could provide a non-invasive and relatively inexpensive tool for identification of such bio-markers. In this study the investigators will use high-density electroencephalographic (EEG) recordings, in order to develop a platform of sensitive and reliable bio-markers for disease progression and response to MR-guided Focused ultrasound thalamotomy (FUS-T) intervention for tremor.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disease the neurochemical hallmark of which is dopamine deficiency in nigrostriatal pathways, and characterized clinically by a movement disorder consisting of rest tremor, bradykinesia, rigidity, impairment of postural reflexes and gait difficulties. The disease may leads to severe neurological dysfunction within several years.

Essential tremor (ET) is a neurological disorder characterized by the presence of action tremor in different body parts mainly in the hands, head, larynx (voice box), tongue, and chin. The lower body is rarely affected.

INSIGHTEC uses MR guided Focused Ultrasound to perform a "non-invasive" thalamotomy to relieve medication refractory tremor in patients with ET or tremor-dominant PD. The effect of MRgFUS is based on tissue destruction targeted to the Vim nucleus of the thalamus which enables a highly accurate and controlled thermal effect.

Ultrasound energy is delivered across the skull, without an incision or craniotomy, heating the targeted tissue above the protein denaturation threshold at temperatures near 60°C. Prior to the delivery of high temperatures, destructive sonication delivery of lower energy focused ultrasound allows for proper anatomic localization, as well as physiologic evaluation of symptom relief and/or any unwanted side effects. This process allows for adjustments before making a permanent lesion. Treatment effects are immediate and the several hour treatment is generally well tolerated with mild sedatives.

The FUS-T procedure was shown as an efficacious procedure for tremor in both ET patients and PD patients; Elminda developed an algorithm of Brain network activation (BNA) Mapping Functional Networks of Brain Activity Using EEG.

Studying brain morphology and function with Neuroimaging and electrophysiological measures is critical for our understanding of the pathology and pathophysiology of PD and ET.

The BNA network can shed a lite on the brain connectivity changes that occur as a result treatment in neurological patients, in this case patients with either PD or ET tremor going through FUS-T.

BNA can help understanding the effects of FUS-T on the brain physiology and perhaps to identify biomarkers that may serve as tools for chosing the best candidates for this treatemnt and optimal treatment parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential Tremor and unilateral tremor-dominant Idiopathic Parkinson's Disease -undergoing ExAblate 4000 Transcranial MR guided focused ultrasound (TcMRgFUS) thalamotomy).

Exclusion Criteria:

* In the investigator's opinion, any unstable or clinically significant condition that would impair the participants' ability to comply with study requirements.
* Patients with significant psychiatric symptoms or history
* Treatment with neuroleptics.
* Currently with lice or open wounds on scalp.
* Significant sensory deficits, e.g., deafness or blindness
* Current drug abuse or alcoholism.
* Pregnancy or not using a reliable method of birth control

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 50 patients with idiopathic PD with tremor 50 patients with Essential tremor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
EEG/ ERP recordings | 2 years
  EEG/ERP: Quantitative EEG based on 64 channel acquisition will be performed during the stimulation treatment to search for discriminatory markers of response to stimulation. Sessions will initially comprise a series of both task (evoked potentials/event-related potentials (ERPs, to be determined) and rest states. The task state will principally be evaluated for brain network analysis (BNA, ElMindA, Israel).

SECONDARY OUTCOMES:
computerized gait analysis | 2 years
  Another optional monitoring procedure is a computerized gait analysis of the Mon4t system (iPhone4, Apple®, Cupertino, California, USA): In order to capture the subject position and motion the investigators will use a standard smartphone. Gait will be assessed by the use of a set of wearable accelerometers, gyroscopes and magnetometers which are all included into the smartphone.